CLINICAL TRIAL: NCT02741102
Title: Uterine Transplant in Absolute Uterine Infertility (AUIF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Stefan G Tullius, Chief , Division of Transplant Surgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P002552
Record Dates: First submitted 2016-02-22; First posted 2016-04-18 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Female Infertility
Keywords: Infertility; AUFI
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Women with AUFI (Experimental): Women with AUFI must meet criteria for uterine transplant. In vitro fertilization to obtain 6 (screened) healthy embryos for cryo-preservation precedes uterine transplant from an appropriate donor The recipient will be required to take potent anti rejection medications including Thymoglobulin, Prednisone, Tacrolimus, Mycophenolate Mofetil (MMF) , later substituted with Azathioprine to avoid birth defects. One year later, up to 6 attempts using 1 screened embryo at a time will be tried to achieve pregnancy. During pregnancy, the high risk pregnancy and transplant teams will follow the recipient. The goal is a full term baby and delivery will be by Caesarian section. A second pregnancy may be attempted. Afterward, the uterus will be explanted.
  Interventions: Procedure: Uterine Transplant

INTERVENTIONS:
Procedure: Uterine Transplant — Treating Absolute Uterine Factor Infertility by Uterus Transplant. Potential recipients undergo IVF to obtain 6 embryos for cryopreservation followed by live donor uterine transplant. After 1 year, embryo transfer is done to achieve pregnancy. Delivery is by Caesarian section. The recipient may have up to 2 children by these methods and then the uterus is removed so that immunosuppression can be stopped.

SUMMARY:
This study will examine the feasibility of initiating a uterine transplant program for Absolute Uterine Factor Infertility (AUFI) at Brigham and Women's Hospital. The investigators plan to screen 30 patients with a goal of enrolling 10 patients. (5 donors and 5 recipients) After careful screening, appropriate candidates will undergo IVF, Uterine Transplantation, Embryo Transfer, Pregnancy and Delivery. Once the uterus is explanted, five years of follow-up is planned.

DETAILED DESCRIPTION:
There are approximately 9.5 million women in the United States with Absolute Uterine Factor Infertility (AUFI).Congenital uterine infertility in women is linked to a malformed or absent mullerian system termed MRKH - Rokitansky's or Mayer-Rokitansky-Kuster-Hauser Syndrome). Additional causes of acquired uterine infertility include a hysterectomy subsequent to life-threatening hemorrhage during childbirth or as a consequence to a hysterectomy related to cervical cancer or for large symptomatic fibroids. Additional causes may include intrauterine adhesions subsequent to surgical abortion or infection.

Uterine transplantation will provide a much needed medical option for many women in the U.S. and overseas who are unable to carry their own children based on uterine infertility. Centers outside of the US have initiated uterus transplant programs. Initial attempts were reported from Saudi Arabia. While the deceased donor transplant had been successful, successful pregnancies were not achieved. Another deceased donor transplant had been performed in Turkey with a uterus procured from a deceased donor. Although several IVF attempts had been performed, they had not resulted in live births.

Uterus transplants from live donors have been successful. In October 2014, Swedish doctors treating a woman born without a uterus, announced the world's first live birth of a healthy baby boy after a live donor uterine transplantation. Since then, an additional three babies have been born in Sweden to mothers who received live donor uterus transplants. A fifth baby is at term and a 6th pregnancy has been reported.

For this study, the investigators plan to screen 30 patients in order to enroll 10 patients, 5 recipients and their respective donors. Prospective recipients will undergo comprehensive medical and psychological evaluation. If deemed an appropriate candidate, In Vitro Fertilization would be started with the goal of obtaining 6 normal embryos for implantation. The uterus of a suitable live donor would then transplanted into the recipient. The recipient would need to take potent anti-rejection drugs and undergo regular assessments for rejection. After one year, embryo transfer to the transplanted uterus would be tried. Up to 6 cycles would be attempted hopefully resulting in pregnancy. If pregnancy results, the recipient would be followed by the high risk pregnancy team. Delivery will be by Caesarian Section. A woman may have up to 2 pregnancies with the transplanted uterus. The uterus is later removed so the recipient no longer has to take anti-rejection drugs.

ELIGIBILITY:
Uterine Transplant Inclusion/Exclusion Criteria

RECIPIENT:Inclusion Criteria

* Age 18-40
* Clinical evidence of AUFI (Absolute Uterine Factor Infertility)
* Able to produce at least 6 normal embryos by IVF for future use
* Reasonable weight with BMI (Body Mass Index) less than 30.
* Normal kidney function
* Able to undergo transplant and be compliant with treatment
* Has stable partner and social supports
* Partner willing to undergo psychological evaluation and receive immunizations as recommended
* Stable home environment to support a child

Exclusion Criteria :

* Active smoking, alcohol use or use of illicit drugs
* Inability to comply with required treatment (taking pills, having biopsies, frequent appointments )
* Having a condition that would make pregnancy or taking anti rejection medicines too risky.
* Active infection: Human Immunodeficiency Virus (HIV) , Tuberculosis, Hepatitis B, Hepatitis C
* History of extensive abdominal or pelvic surgery
* History of abnormal Papanicolaou test (PAP smear) or genital warts
* History of pelvic inflammatory disease

DONOR:Inclusion criteria

* Age over 40 up to age 60
* Has completed having a family
* Previous pregnancies were carried to term (no miscarriages)
* Able to take a birth control pill containing estrogen
* Weight reasonable with BMI (Body Mass Index) of 30 or less
* Good social supports

Exclusion Criteria:

* Active smoking, alcohol use or use of illicit drugs
* Psychiatric illness
* Cervical or endometrial polyps (growths) or tumors in the uterus muscle
* History of more than 1 Caesarean section
* History of abnormal PAP smear or genital warts
* Internal scarring from extensive abdominal or pelvic surgery
* Hypertension, Coronary artery disease, Chronic Obstructive Lung disease (emphysema) and Diabetes
* Active cancer or incompletely treated cancer
* Active infection including Human Immunodeficiency Disease (HIV) , Tuberculosis, Hepatitis B or Hepatitis C
* Significant history of either blood clots or bleeding tendencies
* Evidence of coercion or exchange of money or goods for donating the organ

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-06 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Number of successful live births following uterus transplant/embryo transfer | 2 years after uterine transplant
  Full term live birth by caesarian section after uterus transplant and IVF

SECONDARY OUTCOMES:
Rate of complications during pregnancy in uterus transplant recipient | 9 months after pregnancy achieved by embryo transfer
  Monitoring for pre-eclampsia, hypertension, pre-term delivery
Rate of complications following uterine donation | Up to 2 years post donation
  Monitoring for excessive bleeding , infection and bladder dysfunction
Impact of uterine donation on donor quality of life | Up to 2 years post donation
  Measured by serial SF 36 QOL survey by psychiatrist at pre-donation and at follow-up appointments
Cost comparison for uterine transplant vs. surrogacy vs adoption | Up to 5 years after uterine transplant
  At the end of the study, investigators will calculate average cost of each modality, i.e. transplant vs surrogacy vs adoption to compare the three alternatives to infertility
Impact of uterine transplant on quality of life | Up to 5 years after uterine transplant
  Measured by serial SF 36 QOL survey by psychiatrist pre-transplant and at follow-up appointments..

CONTACTS AND LOCATIONS:
Overall Officials: Stefan G Tullius, M.D., Principal Investigator — Brigham and Womens Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armenti VT, Moritz MJ, Davison JM. Drug safety issues in pregnancy following transplantation and immunosuppression: effects and outcomes. Drug Saf. 1998 Sep;19(3):219-32. doi: 10.2165/00002018-199819030-00005. PMID 9747668
- [Background] Brannstrom M, Johannesson L, Dahm-Kahler P, Enskog A, Molne J, Kvarnstrom N, Diaz-Garcia C, Hanafy A, Lundmark C, Marcickiewicz J, Gabel M, Groth K, Akouri R, Eklind S, Holgersson J, Tzakis A, Olausson M. First clinical uterus transplantation trial: a six-month report. Fertil Steril. 2014 May;101(5):1228-36. doi: 10.1016/j.fertnstert.2014.02.024. Epub 2014 Feb 27. PMID 24582522
- [Background] Christensen, M, Kronberg, CJ, Knudsen UB: Pre-eclampsia and arterial stiffness - a 10 year follow-up of previous pre-eclamptic women. Pregnancy Hyprtens 2015; 5: 72-73.
- [Background] Del Priore G, Saso S, Meslin EM, Tzakis A, Brannstrom M, Clarke A, Vianna R, Sawyer R, Smith JR. Uterine transplantation--a real possibility? The Indianapolis consensus. Hum Reprod. 2013 Feb;28(2):288-91. doi: 10.1093/humrep/des406. Epub 2012 Nov 30. PMID 23202992
- [Background] Josephson MA, McKay DB. Women and transplantation: fertility, sexuality, pregnancy, contraception. Adv Chronic Kidney Dis. 2013 Sep;20(5):433-40. doi: 10.1053/j.ackd.2013.06.005. PMID 23978550
- [Background] Lefkowitz A, Edwards M, Balayla J. The Montreal Criteria for the Ethical Feasibility of Uterine Transplantation. Transpl Int. 2012 Apr;25(4):439-47. doi: 10.1111/j.1432-2277.2012.01438.x. Epub 2012 Feb 23. PMID 22356169
- [Background] Le Ray C, Coulomb A, Elefant E, Frydman R, Audibert F. Mycophenolate mofetil in pregnancy after renal transplantation: a case of major fetal malformations. Obstet Gynecol. 2004 May;103(5 Pt 2):1091-4. doi: 10.1097/01.AOG.0000124986.32858.ba. PMID 15121619
- [Background] McKay DB, Josephson MA. Pregnancy in recipients of solid organs--effects on mother and child. N Engl J Med. 2006 Mar 23;354(12):1281-93. doi: 10.1056/NEJMra050431. No abstract available. PMID 16554530
- [Background] Brannstrom M, Wranning CA, Altchek A. Experimental uterus transplantation. Hum Reprod Update. 2010 May-Jun;16(3):329-45. doi: 10.1093/humupd/dmp049. Epub 2009 Nov 7. PMID 19897849
- [Background] Szekeres-Bartho J, Csernus V, Hadnagy J, Pacsa AS. Immunosuppressive effect of serum progesterone during pregnancy depends on the progesterone binding capacity of the lymphocytes. J Reprod Immunol. 1983 Mar;5(2):81-8. doi: 10.1016/0165-0378(83)90003-7. PMID 6132996
- [Result] Balayla J, Dahdouh EM, Lefkowitz A; Montreal Criteria for the Ethical Feasibility of Uterine Transplantation Research Group. Livebirth after uterus transplantation. Lancet. 2015 Jun 13;385(9985):2351-2. doi: 10.1016/S0140-6736(15)61096-0. No abstract available. PMID 26088636